CLINICAL TRIAL: NCT04180618
Title: Multi-centered Study to Evaluate Patient Satisfaction and Work Efficiency of Medical Staff When Using Personal Health Wallet Service for Emergency Situation
Brief Title: Study to Evaluate Satisfaction Using Personal Health Wallet Service
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2019-07-066-006
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Emergencies
MeSH Terms: conditions — Emergencies | interventions — Emergency Service, Hospital

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients(Care givers) (Experimental): 1. 1,000 patients(caregivers) are enrolled and use the personal health wallet service.
  2. They fill out questionnaire to evaluate the service
  3. Some of them are invited for an in-depth interview.
  Interventions: Other: Personal health wallet service for emergency situation
- Medical staffs (Experimental): 1. 12 medical staffs are enrolled and use the personal health wallet service.
  2. After that, they are invited for an in-depth interview.
  Interventions: Other: Personal health wallet service for emergency situation

INTERVENTIONS:
Other: Personal health wallet service for emergency situation — Patients(caregivers) and medical staffs will be provided the personal health wallet service and evaluate the effectiveness and satisfaction for the service.

SUMMARY:
The investigators developed the service showing patient health record altogether which is managed by each hospital separately and recording the patient health information based on mobile application. This study is a multi-centered study involving three hospitals, providing services to patients, care givers and medical staffs. After the participants use this service, the investigators evaluate the effectiveness and satisfaction of this service through questionnaires and in-depth interviews.

DETAILED DESCRIPTION:
* Background: In emergency situations there are difficulties for treatment in that patient health records are not immediately provided because patient information is separately managed by each hospital. Another reason for the difficulty is that if the patients don't know their personal health record, they can't inform medical staffs of it. In addition, the increase of emergency situation of the chronically ill is also problematic. And patients have a growing desire for their health information. In this situation, the investigators developed the service showing patient health record altogether which is managed by each hospital separately and recording the patient health information based on mobile application.
* Objective: This study evaluates the effectiveness and satisfaction of the developed service in the emergency situation
* Design: Mixed method(questionnaires and interview)
* Setting: In the Department of Emergency at the Samsung Medical Center, the Asan Medical Center, the Dong-A Medical Center, and cooperative hospitals
* Enrollment: 1,000 patients(care givers) and about 12 medical staffs
* Intervention

  1. Patients or care givers

     1. 1,000 patients(care givers) are enrolled and use the personal health wallet service.
     2. The participants fill out questionnaire to evaluate the service
     3. Some of them are invited for an in-depth interview.
  2. Medical staffs

     1. About 12 medical staffs are enrolled and use the personal health wallet service.
     2. After that, the medical staffs are invited for an in-depth interview.

ELIGIBILITY:
Inclusion Criteria:

1. SUS-based usability assessment and survey

   * Patient and caregivers of emergency room at Samsung Medical Center
   * Adults over 19 years old.
   * Those who voluntarily agreed to participate in the research
   * Patients who are past the acute period and in stable condition can agree with them
2. Interview

   * Users of the personal health wallet service for emergency situations among patients and caregivers in the emergency room of Samsung Medical Center
   * Medical staffs at Samsung Medical Center and associated hospitals
   * Adults over 19 years old.
   * Those who voluntarily agreed to participate in the research

Exclusion Criteria:

1. SUS-based usability assessment and survey

   * Anyone who disagrees with this study
   * Patients who are not conscious when leaving the emergency room, patients who are not aware of or are not aware of their orientation, patients who are not aware of their level of awareness, or people who are in shock or in deep shutdown situations) (Even in the above cases, caregivers can be included in the clinical trial target if they are present. )
2. Interview

   * Patient is the same as SUS based usability assessment and exclusion criteria for survey participants
   * In the case of medical staffs, those who do not agree with this study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health care for emergency situations | 2 month for enrollment and study
  SUS(System Usability Scale)-based assessment of patients or care givers satisfaction using personal health care for emergency situations. SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. Its score range is 0~100 and the higher the score, the higher the satisfaction level.

SECONDARY OUTCOMES:
A qualitative study on the satisfaction of patients(caregivers) and medical staffs through interviews | 2 month for enrollment and study
  A qualitative study on the satisfaction of patients(caregivers) and medical staffs through interviews

CONTACTS AND LOCATIONS:
Overall Officials: Taerim KIM, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim SM, Kim T, Cha WC, Lee JH, Kwon IH, Choi Y, Kim JS. User Experience of Mobile Personal Health Records for the Emergency Department: Mixed Methods Study. JMIR Mhealth Uhealth. 2020 Dec 15;8(12):e24326. doi: 10.2196/24326. PMID 33320102